CLINICAL TRIAL: NCT03513978
Title: Comparison of the Effects Between Two Multimodal-programs of Exercises on Joint Position Sense, Dynamic Postural Balance and Counter Movement Jump in Male Soccer Players.
Brief Title: Effects of Two Multimodal-programs of Exercises in Male Soccer Players.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Collaborators: Ilustre Colegio Profesional de Fisioterapeutas de la Comunidad de Madrid (Unknown)
Responsible Party: Principal Investigator, Marcos Jose Navarro Santana, Principal Investigator., University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Undefined
Record Dates: First submitted 2018-03-26; First posted 2018-05-02 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Sports Physical Therapy
Keywords: Soccer; Prevention injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IAI Protocol (Experimental): A progressive exercises with transference to sport protocol, oriented to improve the proprioception.
  Interventions: Other: IAI Exercises Protocol
- FIFA 11+ Protocol (Active Comparator): A typical exercises protocol to soccer
  Interventions: Other: FIFA 11+

INTERVENTIONS:
Other: IAI Exercises Protocol — Progressive exercises to improve the strength and propioception of the male soccer players.
  Arms: IAI Protocol
Other: FIFA 11+ — Progressive exercises protocol to prevent injuries in male soccer players which has been created by "FIFA". It is based in different body wieght exercises to improve the neuromuscular control and stabilization.
  Arms: FIFA 11+ Protocol

SUMMARY:
The prevention of injuries has a close relation with the proprioception. In this sense, the proprioception is defined as the information about the corporal and segmental movement, as well as the position of the body and the corporal segments of oneself in the space. Some authors divide the proprioception into kinesthesia and the Joint Position Sense (JPS).

The hypothesis of the study is the implantation of a progressive multimodal exercise protocol with transferences to sport in the trainings of amateur male soccer players in the age range from 18 to 30 years, can decrease the adverse effects of the fatigue during the high intensity activities and its relation with the JPS. Due to the close relation between fatigue and incidence of injuries, the obtaining of positive results could be an important finding for the design of prevention and rehabilitation protocols in soccer.

ELIGIBILITY:
Inclusion Criteria:

* Soccer Players inscribed in Madrid's Soccer Confederation, who have not been sufferd any injury in the last three months and had been trainning regularly in the last six weeks.

Exclusion Criteria:

* Soccer Players who had been suffered any severe injury in the last six months like (1) fracture in the low limb, (2) ACL injury, (3) grade III ankle sprain or (4) any surgical intervention in the low limb.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Joint Position Sense of the knee | Was measured at baseline (realized before the training), post-treatment (six weeks, realized before the training), ten weeks (before the training) and three months (realized before the trainng)
  A digital inclinometer (range measured in degreesº) was used to assess knee Joint Position Sense in a Closed Kinetic Chain using an active modality (athletes actively reached and maintained the knee). The athletes did three trials to the target position. The average of three trials was used to compared with the target position to obtain the absolute error and relative error.
Joint Position Sense of the knee after the training | Was measured at baseline (realized after the training), post-treatment (six weeks, realized after the training) and three months (realized after the trainng)
  A digital inclinometer (range measured in degreesº) was used to assess knee Joint Position Sense in a Closed Kinetic Chain using an active modality (athletes actively reached and maintained the knee). The athletes did three trials to the target position. The average of three trials was used to compared with the target position to obtain the absolute error and relative error.

SECONDARY OUTCOMES:
Fatigue | Was measured at baseline (after the training), post-treatment (six weeks, after the training), and three months (after the training
  The effort perception was measured with Borg Rating of Perceived Exertion Scale (Borg RPE), a 15-point single-item scale ranging from 6 to 20 (with anchors ranging from 6 "No exertion" to 20 "Maximum exertion") (little or no effort) to 20 (maximun exertion) scores
Lateral Step Down Test | Was measured at baseline (realized before and after the training), post-treatment (six weeks, realized before and after the training), ten weeks (realized only before the training) and three months (realized before and after the training
  Five consecutive test repetitions were then performed. The examiner were positioned 3 m in front of the subject during the test. The examiner evaluated the performance of the test simultaneously and scored the test on a 6-point scale (0-5), according to the criteria outlined by Piva et al. A total score of 0 to 1 was classified as "good" quality of movement, a total score of 2 to 3 was classified as "moderate" quality of movement, and a total score of 4 to 5 was classified as "poor" quality of movement.
Counter movement jump | Was measured at baseline (realized before and after the training), post-treatment (six weeks, realized before and after the training), ten weeks (realized only before the training) and three months (realized before and after the training
  Measured by app "My Jump 2", participants performed each CMJ with hands on their hips, starting from a static standing position and with their legs straight during the flight phase of the jump. The landing was performed simultaneously with either feet keeping ankle dorsiflexion. Participants were instructed to jump as high as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Jose Navarro Santana, MSc, Principal Investigator — Alcala University
Locations (1):
- Plaza de los Irlandeses, Nº 12, 2º C, Alcalá de Henares, Madrid, Spain